CLINICAL TRIAL: NCT07138391
Title: The Efficacy of Chamomile Gummies on Dental Anxiety in Children A Randomized Clinical Trial
Brief Title: Chamomile Gummies and Pediatric Dental Anxiety
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec IR/052502
Record Dates: First submitted 2025-07-05; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; chamomile; children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group will receive one chamomile gummy to chew approximately 30 minutes prior to their dental appointment. The gummy used in this study was Zarbee's Gentle Bedtime Gummies for Kids (Zarbee's Inc., USA).
  Interventions: Drug: chamomile gummy
- The control group (Placebo Comparator): The control group will receive a multivitamin gummy, as a placebo, administered at the same time point (30 minutes prior to the appointment)
  Interventions: Dietary Supplement: a multivitamin gummy

INTERVENTIONS:
Drug: chamomile gummy — The chamomile gummy used in this study was Zarbee's Gentle Bedtime Gummies for Kids (Zarbee's Inc., USA).
  Arms: intervention group
Dietary Supplement: a multivitamin gummy — multivitamins gummies for kids
  Arms: The control group

SUMMARY:
The aim of this study is to evaluate the effect of oral chamomile on reducing dental anxiety in children. Anxiety assessments will be done by recording the pulse rate and blood pressure and by using modified child dental anxiety scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients exhibiting Frankl's behavior rating grade III or IV.
* Children requiring invasive dental treatment in their primary teeth

Exclusion Criteria:

1. Patients with severe dental symptoms (e.g. spontaneous pain, pain not relieved by analgesics).
2. History of allergy to local anesthesia
3. Children who currently use any medication

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of anxiety | 1st measurement before gummy chewing and swallowing 2nd measurement 30 mins after gummy swallowing 3rd measurement after local anesthesia injection 4th measurement after completion of dental work one dental visit
  Anxiety assessments will be done using:
  1) The pulse rate: Pulse rate will be measured using a finger-base type pulse oximeter (Beurer, Ulm, Germany). The children will be asked not to move their hand while the finger pulse oximeter is attached to their left index finger.
Assessment of anxiety | 1st measurement before gummy chewing and swallowing 2nd measurement 30 mins after gummy swallowing 3rd measurement after local anesthesia injection 4th measurement after completion of dental work one dental visit
  Anxiety assessments will be done using:
  2) Blood pressure: this will be measured using a digital blood pressure scale.
Assessment of anxiety | 1st measurement before gummy chewing and swallowing 2nd measurement 30 mins after gummy swallowing 3rd measurement after local anesthesia injection 4th measurement after completion of dental work one dental visit
  Anxiety assessments will be done using:
  3) Modified Child Dental Anxiety Scale:

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No